CLINICAL TRIAL: NCT05492578
Title: A Long-term Extension Study to Evaluate the Long-term Safety, Tolerability and Efficacy of Subcutaneous Amlitelimab in Participants of Previous Amlitelimab Clinical Trials in Moderate to Severe Atopic Dermatitis.
Brief Title: Long-Term Safety and Efficacy Evaluation of Amlitelimab in Participants of Previous Amlitelimab Moderate to Severe Atopic Dermatitis Clinical Trials
Acronym: RIVER-AD
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTS17367; U1111-1269-6490 (Registry Identifier: ICTRP); 2023-506548-18 (Registry Identifier: CTIS); KY1005-CT06 (Other: Sanofi Identifier); 2021-002344-73 (EudraCT Number)
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Adrenal Cortex Hormones; Calcineurin Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Amlitelimab dose level 1 (Experimental): Subcutaneous injection as per protocol
  Interventions: Drug: Amlitelimab; Drug: Topical corticosteroids; Drug: Topical calcineurin inhibitors; Drug: Oral corticosteroids
- Amlitelimab dose level 2 (Experimental): Subcutaneous injection as per protocol
  Interventions: Drug: Amlitelimab; Drug: Topical corticosteroids; Drug: Topical calcineurin inhibitors; Drug: Oral corticosteroids

INTERVENTIONS:
Drug: Amlitelimab — Pharmaceutical form: Solution for injection Route of administration: Subcutaneous
  Other Names: SAR445229
Drug: Topical corticosteroids — Pharmaceutical form: Topical Route of administration: Topical
Drug: Topical calcineurin inhibitors — Pharmaceutical form: Topical Route of administration: Topical
Drug: Oral corticosteroids — Pharmaceutical form: Oral Route of administration: Oral

SUMMARY:
This is an open-label, Phase 2/Phase 3, long-term extension study for treatment of participants of previous amlitelimab clinical trials in moderate to severe atopic dermatitis.

The purpose of this study is to characterize the safety and efficacy of amlitelimab in treated participants with moderate to severe atopic dermatitis (AD) who have previously been enrolled in an amlitelimab clinical trial. All participants will have visits during the treatment period every 4 weeks. Responder participants rolling over from EFC17599 and EFC17600, and responder participants enrolling through screening from DRI17366 will be initiated into drug withdrawal (with no drug administration) at LTS17367 baseline visit to monitor durability of treatment response. If these responder participants relapse during LTS17367, they will have treatment restored. Non-responder participants rolling over from EFC17599 or EFC17600, and non-responder participants enrolling through screening from DRI17366 will have treatment administration from LTS17367 baseline. Participants rolling over from DRI17366, SFY17915 and INT18404 will also have treatment administration from LTS17367 baseline.

Remote visits with home dosing are allowed for the purpose of study drug administration, when applicable. In the case of remote visit with home dosing, the participant or a caregiver may administer study drug after appropriate training. Alternatively, if needed, and based on the investigator's judgement, home visits with healthcare professional assistance or on-site study drug administration visits can be performed. Where participants discontinue amlitelimab permanently during LTS17367, safety follow up will be performed for a minimum of 140 days from the last amlitelimab administration.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 12 years of age inclusive at the time of signing the informed consent.
* Participated in an amlitelimab clinical trial for moderate to severe AD and received study treatment, adequately completed the assessments required for the treatment period.

  * Have reached the rollover timepoint to LTS17367 at the last visit of the treatment period of their feeder study SFY17915, INT18404, EFC17599, or EFC17600
  * Participants in DRI17366 must only be enrolled from 1 of the following 3 groups:

    * The first group: participants at Week 24 in the DRI17336 study who have not achieved an ≥ Eczema Area and Skin Severity Index (EASI)-75 and are Investigator Global Assessment (IGA) ≥ 2.
    * The second group: participants entering LTS17367 between Week 28 and Week 52 of the feeder study, due to loss of clinical response in the part 2 of the feeder study. Timepoints for entering LTS17367 are Weeks 28, 32, 36, 40, 44, 48 or 52.
    * The third group: participants at Week 24 in DRI17366 who have been re-randomized and who subsequently complete the study to Week 52, enter safety follow-up and experience worsening of their AD during safety follow-up.
  * Participated in DRI17366 completing the previous study safety follow up (Week 68) and wish to re-initiate treatment with amlitelimab up to one year after the last visit
* Complied with the previous clinical trial protocol to the satisfaction of the investigator
* Body weight must be ≥25 kg
* Provided signed informed assent/or consent and able to comply with the requirements of the protocol Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Developed a medical condition that would preclude participation as described in the section for permanent discontinuation of the feeder study or LTS17367 protocol
* Known history of or suspected current significant immunosuppression, including history of invasive opportunistic infections or helminthic infections despite infection resolution or otherwise recurrent infections of abnormal frequency or prolonged duration
* History of solid organ or stem cell transplant
* Any malignancies or history of malignancies prior to baseline (except for non-melanoma skin cancer that has been excised and completely cured for more than 5 years prior to baseline)
* Participants positive for human immunodeficiency virus (HIV); participants with any of the following results at Screening (Visit 1) or at any point during the feeder study: presence of HBsAg with or without HBV DNA PCR test, or presence of anti-HBc Ab or presence of anti-HBs Ab with positive HBV DNA PCR test; positive HCVAb confirmed by positive HCV RNA PCR test
* History (within last 2 years prior to baseline) of prescription drug or substance abuse, including alcohol, considered significant by the Investigator
* Participants with active TB, latent TB, a history of incompletely treated TB, suspected extrapulmonary TB infection, non-TB mycobacterial infection, or who are at high risk of contracting TB (such as close contact with individuals with active or latent TB) or received Bacillus Calmette-Guérin (BCG)-vaccination within 12 weeks prior to screening
* Participants with an indeterminate or a confirmed positive IGRA test are excluded from the study unless all of the following conditions are met:

  1. Have a history of prior documented completed chemoprophylaxis for latent TB infection (with a treatment regimen as per local guidelines), OR treated for active TB infection
  2. Have been in written form approved for participation in the present trial by a TB specialist who ruled out latent or active TB infection or other mycobacterial infection in the participant
  3. For whom review and approval from Sponsor have been granted are eligible
* Severe concomitant illness that would in the Investigator's opinion inhibit the participant's participation in the study, including for example, but not limited to, hypertension, renal disease, neurological conditions, heart failure and pulmonary disease
* Skin co-morbidity that would adversely affect the ability to undertake AD assessments (e.g., psoriasis, tinea corporis, lupus erythematosus) as per Investigator's judgment
* Any medical condition which, in the opinion of the Investigator may present an unreasonable risk to the study participant as a result of his/her participation in this clinical study, may make participant's participation unreliable, or may interfere with study assessments
* In the Investigator's opinion, medical conditions related to prior AD medications that have not healed/fully recovered for more than 2 weeks before screening visit, including, but not limited to, conjunctivitis, keratitis, eosinophilic conditions, arthralgia, herpes zoster, thrombosis

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1663 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2029-01-22 (Estimated); Study Completion 2029-01-22 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who experienced treatment-emergent adverse event (TEAE) | Baseline to Week 332

SECONDARY OUTCOMES:
Percentage of participants who experienced treatment-emergent serious adverse events (SAEs) | Baseline to Week 332
Percentage of participants who experienced treatment-emergent adverse events of special interest (AESI) | Baseline to Week 332
Percentage of participants who experienced TEAE leading to treatment discontinuation | Baseline to Week 332
Absolute change from DRI17366 baseline in EASI score at each LTS17367 visit in participants entering the study from DRI17366 Week 24 | DRI17366 Baseline to Week 332
  EASI measures the severity & extent of AD based on 4 AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation] & lichenification). Total score ranges from 0 (minimum) to 72 (maximum), higher scores indicated greater severity of AD.
Percent change from DRI17366 baseline in EASI score at each LTS17367 visit in participants entering the study from DRI17366 Week 24 | DRI17366 Baseline to Week 332
  EASI measures the severity & extent of AD based on 4 AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation] & lichenification). Total score ranges from 0 (minimum) to 72 (maximum), higher scores indicated greater severity of AD.
Proportion of participants with EASI50/EASI75/EASI90/EASI100 from DRI17366 baseline at each LTS17367 visit in participants entering the study from DRI17366 Week 24 | DRI17366 Baseline to Week 332
  EASI measures the severity & extent of AD based on 4 AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation] & lichenification). Total score ranges from 0 (minimum) to 72 (maximum), higher scores indicated greater severity of AD. EASI50: >= 50% reduction in score from baseline; EASI75: >= 75% reduction in score from baseline; EASI90: >= 90% reduction in score from baseline; EASI100: >= 100% reduction in score from baseline.
Proportion of participants with a response of Validated Investigator Global Assessment scale for atopic dermatitis (vIGA-AD) 0 or 1 at each LTS17367 visit in participants entering the study from DRI17366 Week 24 | Baseline to Week 332
  The vIGA-AD is an assessment instrument used to rate the severity of AD globally, based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), higher score indicated higher severity.
Proportion of participants with vIGA-AD score 0/1 in all participants entering the study [each LTS17367 visit] | Baseline to Week 332
  The vIGA-AD is an assessment instrument used to rate the severity of AD globally, based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), higher score indicated higher severity.
Proportion of participants with vIGA-AD score 0 [each LTS17367 visit] | Baseline to Week 332
  The vIGA-AD is an assessment instrument used to rate the severity of AD globally, based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), higher score indicated higher severity.
Proportion of participants with vIGA-AD score 0 or 1 with presence of only barely perceptible erythema (no induration/papulation, no lichenification, no oozing or crusting) at each LTS17367 visit | Baseline to Week 332
  The vIGA-AD is an assessment instrument used to rate the severity of AD globally, based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), higher score indicated higher severity.
Time to first vIGA-AD 0/1 after LTS17367 enrollment in those participants who had not achieved vIGA-AD 0/1 by the time of LTS17367 enrollment | Baseline to Week 332
  The vIGA-AD is an assessment instrument used to rate the severity of AD globally, based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), higher score indicated higher severity.
Absolute change from feeder study baseline in EASI score in all participants entering the study [each LTS17367 visit] | Baseline to Week 332
  EASI measures the severity & extent of AD based on 4 AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation] & lichenification). Total score ranges from 0 (minimum) to 72 (maximum), higher scores indicated greater severity of AD.
Percent change from feeder study baseline in EASI score in all participants entering the study [each LTS17367 visit] | Baseline to Week 332
  EASI measures the severity & extent of AD based on 4 AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation] & lichenification). Total score ranges from 0 (minimum) to 72 (maximum), higher scores indicated greater severity of AD.
Proportion of participants with EASI50/EASI75/EASI90 in all participants entering the study [each LTS17367 visit] | Baseline to Week 332
  EASI measures the severity & extent of AD based on 4 AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation] & lichenification). Total score ranges from 0 (minimum) to 72 (maximum), higher scores indicated greater severity of AD. EASI50: >= 50% reduction in score from baseline; EASI75: >= 75% reduction in score from baseline; EASI90: >= 90% reduction in score from baseline.
Time to first EASI75/EASI90 in those participants who had not achieved it by the time of LTS17367 enrollment | Baseline to Week 332
  EASI measures the severity & extent of AD based on 4 AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation] & lichenification). Total score ranges from 0 (minimum) to 72 (maximum), higher scores indicated greater severity of AD. EASI75: >= 75% reduction in score from baseline; EASI90: >= 90% reduction in score from baseline.
Proportion of participants requiring topical treatment in all participants entering the study [each LTS17367 visit] | Baseline to Week 332
Proportion of participants requiring rescue treatment [each LTS17367 visit]: all treatments in all participants entering the study | Baseline to Week 332
Number of days on topical medication (per patient-year) in all participants entering the study | Baseline to Week 332
Change from feeder study baseline atopic dermatitis control tool (ADCT) in all participants entering the study [each LTS17367 visit] | Baseline to Week 332
  ADCT is a six-item patient self-administered instrument designed and validated to assess atopic dermatitis (AD) control. The score ranges from 0-24 with higher scores indicate worsening disease control.
Change from feeder study baseline in dermatology life quality index (DLQI/cDLQI) in all participants entering the study [each LTS17367 visit] | Baseline to Week 332
  The DLQI is a validated 10-item questionnaire to measure dermatology specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
  The children's DLQI (cDLQI) measures dermatology specific quality of life (QoL) in children patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Change from feeder study baseline in patient oriented eczema measure (POEM) in all participants entering the study [each LTS17367 visit] | Baseline to Week 332
  The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms on a scale ranging from 0 to 4 (0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, 4 = all days). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (severe disease). Higher scores indicated more severe disease and poor quality of life.
Change from feeder study baseline in body surface area affected by AD (BSA-AD) [each LTS17367 visit] | Baseline to Week 332
  BSA-AD measured as percentage of body affected by AD.
Time from enrollment in LTS17367 to first loss of vIGA-AD 0 in those participants who were vIGA-AD 0 at LTS17367 rollover from EFC17600 (ESTUARY) and EFC17599 (AQUA) | Baseline to Week 332
  The vIGA-AD is an assessment instrument used to rate the severity of AD globally, based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), higher score indicated higher severity.
Time from enrollment in LTS17367 to first loss EASI75 in those participants who had reached EASI75 at LTS17367 rollover coming from EFC17600 (ESTUARY) and EFC17599 (AQUA) | Baseline to Week 332
  EASI measures the severity & extent of AD based on 4 AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation] & lichenification). Total score ranges from 0 (minimum) to 72 (maximum), higher indicated greater severity of AD. EASI75: >= 75% reduction in score from baseline.
Time from enrollment in LTS17367 to first loss of vIGA-AD 0/1 in those participants who were vIGA-AD 0/1 at LTS17367 rollover from EFC17600 (ESTUARY) and EFC17599 (AQUA) | Baseline to Week 332
  The vIGA-AD is an assessment instrument used to rate the severity of AD globally, based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), higher score indicated higher severity.
Time from LTS17367 baseline to re-treatment with amlitelimab in those participants who were vIGA-AD 0/1 at LTS17367 rollover from EFC17600 (ESTUARY) and EFC17599 (AQUA) | Baseline to Week 332
  The vIGA-AD is an assessment instrument used to rate the severity of AD globally, based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2
  = mild; 3 = moderate; 4 = severe), higher score indicated higher severity.
Time from last amlitelimab dose in feeder study to re-treatment with amlitelimab in those participants who were vIGA-AD 0/1 at LTS17367 rollover from EFC17600 (ESTUARY) and EFC17599 (AQUA) | Baseline to Week 332
  The vIGA-AD is an assessment instrument used to rate the severity of AD globally, based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2
  = mild; 3 = moderate; 4 = severe), higher score indicated higher severity.
Serum amlitelimab concentration assessed at prespecified time points through the end of the study | Baseline to Week 332
  Serum amlitelimab concentration assessed at prespecified time points through the end of the study.
Number of participants with anti-drug antibodies (ADAs) of amlitelimab at specified timepoints | Baseline to Week 332

CONTACTS AND LOCATIONS:
Locations (281):
- United States (69):
  - Allervie Clinical Research - Birmingham- Site Number : 8401101, Birmingham, Alabama
  - Cahaba Dermatology & Skin Health Center- Site Number : 8401066, Birmingham, Alabama
  - Center for Dermatology and Plastic Surgery- Site Number : 8401119, Scottsdale, Arizona
  - Scottsdale Clinical Trials- Site Number : 8401149, Scottsdale, Arizona
  - Arkansas Research Trials- Site Number : 8401244, North Little Rock, Arkansas
  - Orange County Clinical Trials- Site Number : 8401271, Anaheim, California
  - Encino Research Center- Site Number : 8401042, Encino, California
  - First OC Dermatology- Site Number : 8401025, Fountain Valley, California
  - Center for Dermatology Clinical Research- Site Number : 8401018, Fremont, California
  - Sunwise Clinical Research- Site Number : 8401022, Lafayette, California
  - Antelope Valley Clinical Trials- Site Number : 8401099, Lancaster, California
  - Torrance Clinical Research - Narbonne Avenue- Site Number : 8401027, Lomita, California
  - Long Beach Clinical Trials- Site Number : 8401188, Long Beach, California
  - Dermatology Research Associates - Los Angeles- Site Number : 8401092, Los Angeles, California
  - LA Universal Research Center- Site Number : 8401064, Los Angeles, California
  - Cura Clinical Research - Oxnard- Site Number : 8401142, Oxnard, California
  - Southern California Dermatology- Site Number : 8401043, Santa Ana, California
  - Clinical Science Institute- Site Number : 8401028, Santa Monica, California
  - Paradigm Clinical Research - Wheat Ridge- Site Number : 8401245, Wheat Ridge, Colorado
  - Encore Medical Research of Boynton Beach- Site Number : 8401030, Boynton Beach, Florida
  - St. Jude Clinical Research- Site Number : 8401287, Doral, Florida
  - Alliance for Multispeciality Research - Fort Myers- Site Number : 8401111, Fort Myers, Florida
  - Direct Helpers Research Center- Site Number : 8401056, Hialeah, Florida
  - Doral Medical Research - Hialeah- Site Number : 8401094, Hialeah, Florida
  - Clever Medical Research- Site Number : 8401160, Miami, Florida
  - Medical Research Center of Miami II- Site Number : 8401019, Miami, Florida
  - Acevedo Clinical Research Associates- Site Number : 8401088, Miami, Florida
  - Sanchez Clinical Research- Site Number : 8401095, Miami, Florida
  - Future Care Solution - Miami- Site Number : 8401144, Miami, Florida
  - Florida International Research Center- Site Number : 8401091, Miami, Florida
  - Savin Medical Group - Miami Lakes- Site Number : 8401085, Miami Lakes, Florida
  - Wellness Clinical Research - Miami Lakes - 8181 Northwest 154th Street- Site Number : 8401109, Miami Lakes, Florida
  - K2 South Orlando - South Orange Avenue- Site Number : 8401268, Orlando, Florida
  - Global Clinical Professionals (GCP)- Site Number : 8401045, St. Petersburg, Florida
  - Clinical Research Trials of Florida- Site Number : 8401023, Tampa, Florida
  - Alliance Clinical Research of Tampa- Site Number : 8401013, Tampa, Florida
  - First Georgia Physician Group- Site Number : 8401190, Fayetteville, Georgia
  - Aeroallergy Research Laboratory- Site Number : 8401004, Savannah, Georgia
  - Northwestern University- Site Number : 8401038, Chicago, Illinois
  - Equity Medical - Bowling Green- Site Number : 8401296, Bowling Green, Kentucky
  - Skin Sciences- Site Number : 8401039, Louisville, Kentucky
  - Velocity Clinical Research at The Dermatology Clinic - Baton Rouge- Site Number : 8401072, Baton Rouge, Louisiana
  - MedPharmics - Covington- Site Number : 8401137, Covington, Louisiana
  - BRCR Global Gretna- Site Number : 8401243, Gretna, Louisiana
  - Revival Research Institute - Troy- Site Number : 8401012, Troy, Michigan
  - Oakland Medical Center- Site Number : 8401116, Troy, Michigan
  - Allergy & Immunology Associates of Ann Arbor- Site Number : 8401078, Ypsilanti, Michigan
  - SKY Integrative Medical Center/SKYCRNG - Ridgeland- Site Number : 8401058, Ridgeland, Mississippi
  - Skin Specialists- Site Number : 8401068, Omaha, Nebraska
  - Pulmonology Group - Henderson- Site Number : 8401169, Henderson, Nevada
  - The University of New Mexico- Site Number : 8401263, Albuquerque, New Mexico
  - Equity Medical- Site Number : 8401239, New York, New York
  - Skin Search Rochester- Site Number : 8401216, Rochester, New York
  - Axis Clinical Trials- Site Number : 8401196, Fargo, North Dakota
  - Best Skin Research - Camp Hill- Site Number : 8401031, Camp Hill, Pennsylvania
  - Paddington Testing Company- Site Number : 8401041, Philadelphia, Pennsylvania
  - Clinical Research of Philadelphia- Site Number : 8401193, Philadelphia, Pennsylvania
  - Dermatology Associates of Plymouth Meeting- Site Number : 8401147, Plymouth Meeting, Pennsylvania
  - Velocity Clinical Research - Columbia- Site Number : 8401176, Columbia, South Carolina
  - Health Concepts - Site Number : 8401059, Rapid City, South Dakota
  - Arlington Research Center- Site Number : 8401248, Arlington, Texas
  - Modern Research Associates- Site Number : 8401093, Dallas, Texas
  - Reveal Research Institute - Dallas- Site Number : 8401219, Dallas, Texas
  - SMS Clinical Research- Site Number : 8401182, Mesquite, Texas
  - Synapse Clinical Research - Missouri City- Site Number : 8401148, Missouri City, Texas
  - Stryde Research - Epiphany Dermatology- Site Number : 8401185, Southlake, Texas
  - Complete Dermatology - Sugar Land- Site Number : 8401061, Sugar Land, Texas
  - Virginia Dermatology & Skin Cancer Center- Site Number : 8401047, Norfolk, Virginia
  - Wyoming Research Foundation- Site Number : 8401234, Cheyenne, Wyoming
- Argentina (13):
  - Investigational Site Number : 0320006, Rosario, Santa Fe Province
  - Investigational Site Number : 0320007, Rosario, Santa Fe Province
  - Investigational Site Number : 0320011, Buenos Aires
  - Investigational Site Number : 0320016, Buenos Aires
  - Investigational Site Number : 0320008, Buenos Aires
  - Investigational Site Number : 0320010, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320009, Buenos Aires
  - Investigational Site Number : 0320019, Buenos Aires
  - Investigational Site Number : 0320005, Buenos Aires
  - Investigational Site Number : 0320014, Córdoba
  - Investigational Site Number : 0320013, Mendoza
- Australia (7):
  - Investigational Site Number : 0360010, Westmead, New South Wales
  - Investigational Site Number : 0360007, Woolloongabba, Queensland
  - Investigational Site Number : 0363002, Carlton, Victoria
  - Investigational Site Number : 0363003, Melbourne, Victoria
  - Investigational Site Number : 0360006, Melbourne, Victoria
  - Investigational Site Number : 0363001, Parkville, Victoria
  - Investigational Site Number : 0361006, Traralgon, Victoria
- Brazil (8):
  - Centro de Pesquisas da Clínica IBIS- Site Number : 0760002, Salvador, Estado de Bahia
  - PUC Trials- Nucleo de Pesquisa clinica da Escola de Medicina da PUCPR- Site Number : 0760023, Curitiba, Paraná
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre- Site Number : 0760005, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina do ABC- Site Number : 0760001, Santo André, São Paulo
  - Clinica de Alergia Martti Antila- Site Number : 0760006, Sorocaba, São Paulo
  - CCBR / IBPClin - Instituto Brasil de Pesquisa Clínica- Site Number : 0760018, Rio de Janeiro
  - Hospital Alemao Oswaldo Cruz - São Paulo- Site Number : 0760010, São Paulo
  - Centro de Desenvolvimento em Estudos ClÌnicos Brasil- Site Number : 0760014, São Paulo
- Bulgaria (5):
  - Investigational Site Number : 1002004, Pleven
  - Investigational Site Number : 1002005, Sofia
  - Investigational Site Number : 1002003, Sofia
  - Investigational Site Number : 1002006, Sofia
  - Investigational Site Number : 1002002, Sofia
- Canada (26):
  - Investigational Site Number : 1240039, Calgary, Alberta
  - Investigational Site Number : 1240019, Calgary, Alberta
  - Investigational Site Number : 1240023, Calgary, Alberta
  - Investigational Site Number : 1240016, Edmonton, Alberta
  - Investigational Site Number : 1240031, Edmonton, Alberta
  - Investigational Site Number : 1240040, Surrey, British Columbia
  - Investigational Site Number : 1240041, Winnipeg, Manitoba
  - Investigational Site Number : 1240033, Ajax, Ontario
  - Investigational Site Number : 1240014, Barrie, Ontario
  - Investigational Site Number : 1240020, Hamilton, Ontario
  - Investigational Site Number : 1240053, London, Ontario
  - Investigational Site Number : 1240017, London, Ontario
  - Investigational Site Number : 1241106, Markham, Ontario
  - Investigational Site Number : 1240018, Newmarket, Ontario
  - Investigational Site Number : 1241108, Niagara Falls, Ontario
  - Investigational Site Number : 1240034, Ottawa, Ontario
  - Investigational Site Number : 1240024, Richmond Hill, Ontario
  - Investigational Site Number : 1240021, Toronto, Ontario
  - Investigational Site Number : 1240012, Toronto, Ontario
  - Investigational Site Number : 1240026, Toronto, Ontario
  - Investigational Site Number: 1240035, Toronto, Ontario
  - Investigational Site Number : 1241107, Waterloo, Ontario
  - Investigational Site Number : 1241101, Windsor, Ontario
  - Investigational Site Number : 1240006, Québec, Quebec
  - Investigational Site Number: 1240028, Regina, Saskatchewan
  - Investigational Site Number : 1240036, Saskatoon, Saskatchewan
- Chile (8):
  - Investigational Site Number : 1520004, Valdivia, Los Ríos Region
  - Investigational Site Number : 1520013, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520008, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520010, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
- China (21):
  - Investigational Site Number : 1560004, Beijing
  - Investigational Site Number : 1560050, Changsha
  - Investigational Site Number : 1560022, Chengdu
  - Investigational Site Number : 1560043, Fuzhou
  - Investigational Site Number : 1560021, Guangzhou
  - Investigational Site Number : 1560025, Guangzhou
  - Investigational Site Number : 1560036, Guangzhou
  - Investigational Site Number : 1560058, Guangzhou
  - Investigational Site Number : 1560044, Hangzhou
  - Investigational Site Number : 1560002, Hangzhou
  - Investigational Site Number : 1560006, Hangzhou
  - Investigational Site Number : 1560029, Hangzhou
  - Investigational Site Number : 1560024, Ningbo
  - Investigational Site Number : 1560035, Ningbo
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560041, Shenyang
  - Investigational Site Number : 1560026, Shenyang
  - Investigational Site Number : 1560023, Wenzhou
  - Investigational Site Number : 1560038, Wuhan
  - Investigational Site Number : 1560003, Wuxi
  - Investigational Site Number : 1560028, Zhenjiang
- Czechia (12):
  - Investigational Site Number : 2032108, Brno
  - Investigational Site Number : 2032106, Kutná Hora
  - Investigational Site Number : 2032105, Nový Jičín
  - Investigational Site Number : 2030010, Olomouc
  - Investigational Site Number : 2032104, Ostrava
  - Investigational Site Number : 2030009, Pilsen
  - Investigational Site Number : 2032102, Prague
  - Investigational Site Number : 2030008, Prague
  - Investigational Site Number : 2032101, Prague
  - Investigational Site Number : 2032103, Prague
  - Investigational Site Number : 2030011, Prague
  - Investigational Site Number : 2030006, Prague
- France (5):
  - Investigational Site Number : 2500008, Antony
  - Investigational Site Number : 2500011, Bordeaux
  - Investigational Site Number : 2500014, Clermont-Ferrand
  - Investigational Site Number : 2500001, Lille
  - Investigational Site Number : 2500012, Rouen
- Germany (9):
  - Investigational Site Number : 2760009, Bad Bentheim
  - Investigational Site Number : 2762203, Berlin
  - Investigational Site Number : 2762202, Blankenfelde-Mahlow
  - Investigational Site Number : 2761001, Dresden
  - Investigational Site Number : 2762207, Gera
  - Investigational Site Number : 2760017, Hamburg
  - Investigational Site Number : 2762208, Kiel
  - Investigational Site Number : 2761002, Lübeck
  - Investigational Site Number : 2762201, Münster
- Investigational Site Number : 3000001, Athens, Greece
- Hungary (2):
  - Investigational Site Number : 3482303, Debrecen
  - Investigational Site Number : 3482306, Szolnok
- Israel (4):
  - Investigational Site Number : 3760005, Beersheba
  - Investigational Site Number : 3760003, Jerusalem
  - Investigational Site Number : 3760007, Tel Aviv
  - Investigational Site Number : 3760008, Tel Litwinsky
- Italy (5):
  - Investigational Site Number : 3800017, Naples, Napoli
  - Investigational Site Number : 3800016, Chieti
  - Investigational Site Number : 3800021, Modena
  - Investigational Site Number : 3800015, Perugia
  - Investigational Site Number : 3800020, Torino
- Japan (20):
  - Investigational Site Number : 3920007, Hiroshima, Hiroshima
  - Investigational Site Number : 3923114, Obihiro-Shi, Hokkaido
  - Investigational Site Number : 3923101, Sapporo, Hokkaido
  - Investigational Site Number : 3920006, Kobe, Hyōgo
  - Investigational Site Number : 3923108, Kagoshima, Kagoshima-ken
  - Investigational Site Number : 3920005, Sagamihara-shi, Kanagawa
  - Investigational Site Number : 3923113, Yokohama, Kanagawa
  - Investigational Site Number : 3920003, Kyoto, Kyoto
  - Investigational Site Number : 3923110, Sakai-shi, Osaka
  - Investigational Site Number : 3920002, Iruma-gun, Saitama
  - Investigational Site Number : 3923106, Shimotsuga-gun, Tochigi
  - Investigational Site Number : 3923112, Adachi-Ku, Tokyo
  - Investigational Site Number : 3923115, Chuo-Ku, Tokyo
  - Investigational Site Number : 3923104, Edogawa-Ku, Tokyo
  - Investigational Site Number : 3923107, Minato-Ku, Tokyo
  - Investigational Site Number : 3923105, Setagaya-Ku, Tokyo
  - Investigational Site Number : 3920001, Tachikawa-shi, Tokyo
  - Investigational Site Number : 3923109, Habikino-shi
  - Investigational Site Number : 3923102, Kyoto
  - Investigational Site Number : 3923113, Yokohama
- Poland (22):
  - Investigational Site Number : 6162407, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6162409, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6162406, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number: 6160010, Tarnów, Lesser Poland Voivodeship
  - Investigational Site Number : 6162414, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6162418, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6162417, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6162415, Lodz, Lódzkie
  - Investigational Site Number : 6162416, Lódz, Lódzkie
  - Investigational Site Number : 6162411, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6162413, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6162401, Rzeszów, Podkarpackie Voivodeship
  - Investigational Site Number : 6162419, Bialystok, Podlaskie Voivodeship
  - Investigational Site Number : 6162403, Gdansk, Pomeranian Voivodeship
  - Investigational Site Number : 6162402, Gdansk, Pomeranian Voivodeship
  - Investigational Site Number : 6160006, Gdansk, Pomeranian Voivodeship
  - Investigational Site Number : 6162404, Gdynia, Pomeranian Voivodeship
  - Investigational Site Number : 6162405, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6162410, Szczecin, West Pomeranian Voivodeship
  - Investigational Site Number : 6162408, Krakow
  - Investigational Site Number : 6160022, Lodz
  - Investigational Site Number : 6162412, Warsaw
- Portugal (3):
  - Investigational Site Number : 6200004, Lisbon
  - Investigational Site Number : 6200001, Lisbon
  - Investigational Site Number : 6200003, Porto
- Investigational Site Number : 6820001, Riyadh, Saudi Arabia
- South Africa (5):
  - Investigational Site Number : 7100015, Benoni
  - Investigational Site Number : 7100010, Cape Town
  - Investigational Site Number: 7100009, Claremont
  - Investigational Site Number : 7100012, Durban
  - Investigational Site Number : 7100001, Durban
- South Korea (11):
  - Investigational Site Number : 4100012, Gwangju, Gwangju
  - Investigational Site Number : 4100002, Ansan-si, Gyeonggi-do
  - Investigational Site Number : 4100009, Suwon, Gyeonggi-do
  - Investigational Site Number : 4100003, Yangsan, Gyeongsangnam-do
  - Investigational Site Number : 4100015, Incheon, Incheon-gwangyeoksi
  - Investigational Site Number : 4100013, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100007, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100010, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100006, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100011, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100008, Daegu
- Spain (8):
  - Investigational Site Number : 7240012, Las Palmas de Gran Canaria, Canary Islands
  - Investigational Site Number : 7240002, Badalona, Catalunya [Cataluña]
  - Investigational Site Number : 7242504, Pontevedra, Galicia [Galicia]
  - Investigational Site Number : 7240023, Burjassot - Valencia, Valenciana, Comunidad
  - Investigational Site Number : 7242505, Alicante
  - Investigational Site Number : 7242501, Córdoba
  - Investigational Site Number : 7240018, Granada
  - Investigational Site Number : 7242503, Madrid
- Taiwan (4):
  - Investigational Site Number : 1583201, Kaohsiung City
  - Investigational Site Number : 1583202, Taichung
  - Investigational Site Number : 1580001, Taipei
  - Investigational Site Number : 1583203, Taoyuan
- Turkey (Türkiye) (3):
  - Investigational Site Number : 7920005, Istanbul
  - Investigational Site Number : 7920004, Kayseri
  - Investigational Site Number : 7920008, Şahinbey
- Investigational Site Number : 7840001, Abu Dhabi, United Arab Emirates
- United Kingdom (8):
  - Investigational Site Number : 8260013, Bristol, Bristol, City of
  - Investigational Site Number : 8260006, Glasgow, Glasgow City
  - Investigational Site Number : 8260003, Portsmouth, Hampshire
  - Investigational Site Number : 8260004, Leicester, Leicestershire
  - Investigational Site Number : 8262603, London, London, City of
  - Investigational Site Number : 8262601, London, London, City of
  - Investigational Site Number : 8260010, Sutton in Ashfield, Nottinghamshire
  - Investigational Site Number : 8260008, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LTS17367 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25304&tenant=MT_SNY_9011